CLINICAL TRIAL: NCT06053593
Title: Ketostix® and Keto-Diastix® Performance Study
Status: Completed | Type: Observational
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: GCA-PRO-2022-002-01
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Testing of Ketostix by Persons with Diabetes.: Each PWD will test Ketostix in their self-collected urine, complete a labeling evaluation, and test four urine control solutions.
  Interventions: Device: Testing of self collected urine; Device: Labeling Evaluation; Device: Urine Control testing
- Testing of Keto-Diastix by Persons with Diabetes.: Each PWD will test Keto-Diastix in their self-collected urine, complete a labeling evaluation, and test four urine control solutions.
  Interventions: Device: Testing of self collected urine; Device: Labeling Evaluation; Device: Urine Control testing

INTERVENTIONS:
Device: Testing of self collected urine — Each PWD will test their self-collected urine.
Device: Labeling Evaluation — Each PWD will complete a labeling evaluation.
Device: Urine Control testing — Each PWD will test four urine control solutions.

SUMMARY:
Persons with Diabetes (PWDs), at minimum of (n=120) will successfully collect their urine and test with two Ascensia strip products. The products are: Ketostix and Keto-Diastix.

DETAILED DESCRIPTION:
Persons with Diabetes (PWDs), at minimum of (n=120) will successfully collect their urine and test with two Ascensia strip products.

1. Demonstrate that untrained PWDs can successfully read the Instructions for Use and use Ketostix and Keto-Diastix reagent strips for Urinalysis with no training. Urine samples from the PWDs will be collected and then tested by the PWD and will be compared to the reference assay results.
2. Demonstrate Ease of Use by PWDs with a Labeling Evaluation Survey for Ketostix and Keto-Diastix reagent strips. Participants will respond to a survey using a 5 point Likert scale with 5= Strongly Agree, 4= Agree, 3=Neutral, 2=Disagree, 3=Strongly Disagree.
3. Demonstrate that persons with diabetes (PWDs) can successfully test urinalysis control solutions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years of age.
* Diagnosed with Diabetes Mellitus (Type 1 or Type 2)
* Able to speak, read and understand English (subjects must demonstrate ability to read a paragraph from the first page of the package insert to qualify for the study).
* Willing to complete all study procedures.

Exclusion Criteria:

* Physical, visual, or neurological impairments that would make the person unable to perform urine collection and testing with the urine strips as determined by the PI.
* Intake of Vitamin C supplements (multi-vitamins are permitted)
* Prior experience testing glucose or ketones in urine with Ketostix and Keto-Diastix Reagent strips.
* Currently taking compounds such as mesna (Mesnex)
* Currently taking any medications containing azo dyes (e.g., Pyridium, Gantrisin, Gantanol), nitrofurantoin (Macrodantin, Furadantin).
* Currently taking medications such as levodopa.
* Working for a medical laboratory, hospital or other clinical setting that involves training in the urinalysis lab or use of urinalysis test strips.
* Working for a competitive medical device company (Urine Strip manufacturer) or having an immediate family member or living with someone who works for such a company.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee on the study form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person with Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Testing of self collected urine | Day 1
  Number of Participants with results from self collected urine that are within one color block of reference analyzer
Labeling evaluation | Day 1
  Number of Participants with Responses that are a 3,4, or 5 on a 5 point Likert Scale.
Testing of Urine controls | Day 1
  Number of Participants with Reponses that read within one color block.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Christenson, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No